CLINICAL TRIAL: NCT05841576
Title: Anaesthetic Management Guided by Cellular Oxygen Metabolism Measurements in Abdominal Surgery: a Randomised Controlled Trial
Brief Title: Anaesthetic Management Guided by COMET Measurements
Acronym: AIMED COMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rick Hulskes (Other)
Collaborators: Photonics Healthcare B.V., Utrecht, The Netherlands (Unknown)
Responsible Party: Sponsor-Investigator, Rick Hulskes, Study coordinator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL77186.018.21; NL9505 (Registry Identifier: Netherlands Trial Register)
Record Dates: First submitted 2022-11-23; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Mitochondrial Oxygenation Measurement; Surgical Site Infection
Keywords: mitochondria; mitochondrial oxygenation; tissue oxygenation; microcirculation; surgical site infection; wound infection; abdominal surgery
MeSH Terms: conditions — Surgical Wound Infection; Wound Infection

STUDY DESIGN:
Intervention Model Description: A randomised, controlled, single-centre, parallel-arm, patient-blinded trial
Who Masked: Participant
Masking Description: The mitoPO2 in the control group is covered and made invisible to the anaesthetists. During the procedure, the outcome assessor is present to troubleshoot the device when needed and is also not blinded. Patients, surgeons and healthcare professionals during the postoperative period are blinded to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COMET monitoring device (Experimental): Anaesthetists for patients allocated to the intervention group were asked to strive and maintain the intraoperative mitoPO2 to the individualised preoperative baseline mitoPO2 with a minimum of 66 mmHg
  Interventions: Other: COMET monitoring device
- Control group (No Intervention): Patients allocated to the control group were treated as per anaesthetist preference and followed our institution's conventional care

INTERVENTIONS:
Other: COMET monitoring device — Cellular Oxygen METabolism (COMET) mitochondrial oxygen tension monitoring device
  Arms: COMET monitoring device

SUMMARY:
Surgical site infection (SSI) is a significant cause of morbidity and mortality, prolonged hospital stays and healthcare costs. Perioperative low tissue oxygen tension is associated with a high risk of SSI. Standard anaesthetic management guided by continuous monitoring of oxygen delivery with a non-invasive method of measuring mitochondrial oxygenation tension (mitoPO2) using the Cellular Oxygen METabolism (COMET) monitor may benefit the intraoperative oxygenation on the tissue level. This randomised, controlled, single-centre, parallel-arm, patient-blinded trial aims to investigate if standard anaesthetic management guided by mitoPO2 monitoring results in higher tissue oxygen tension including patients undergoing elective abdominal surgery. Anaesthetists in the intervention group strive to a minimum mitoPO2 of 66 mmHg. Patients in the control group receive standard care. The primary outcome is the difference in means of the mean mitoPO2 during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients are at least 18 years old
* Patients undergo elective open or laparoscopic abdominal surgery with an expected minimal total incision size of 5 cm
* Patients are able and willing to give written informed consent

Exclusion Criteria:

* Known photodermatoses of varying pathology and frequency
* Mitochondrial disease
* Porphyria
* Skin lesions on the upper arm which impede measurements
* Hypersensitivity to the active substance or the 5-ALA medicated plaster material
* Emergency surgery
* Reoperation for complications from recent surgery (within last three months)
* Participation in another study with interference with this study
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-11-26 (Actual); Study Completion 2022-11-26 (Actual)

PRIMARY OUTCOMES:
Mean mitoPO2 during abdominal surgery over time | during surgery
  Absolute difference between the means of the mean mitoPO2

SECONDARY OUTCOMES:
Surgical site infection | 30 days follow-up
  Surgical site infection rate according to the CDC definition [1].
MitoPO2 above baseline | during surgery
  The percentage of surgery time that the intraoperative mitoPO2 is above baseline
Exploration analysis of the correlation coefficients between the intraoperative mitoPO2 and the intraoperative monitoring measurement values | during intraoperative anaesthetic procedure
  Calculation of the correlation coefficients between the intraoperative mitoPO2 values and the intraoperative values of each monitoring measurement. The measurement pairs are defined as measurements performed within the same time interval. The mean value is used if multiple measurements of the same type have been performed in that time interval. The outcomes are the pooled correlation coefficients of the correlation between the mitoPO2 and each monitoring measure. We going to examine the following monitoring measurements: non-invasive or arterial blood pressure in mmHg, plethysmographic variability index, heart rate, peripheral oxygen saturation, temperature in Celsius, end-tidal oxygen in mmHg, end-tidal carbon dioxide in mmHg and amplitude frequency effect (pulse pressure and heart rate)).
The respective effect per intervention in mitoPO2 after notification in which mitoPO2 aids decision making on anaesthetic management | during intraoperative anaesthetic procedure
  The potential effects of the anaesthetic interventions on the mitoPO2 values is assessed amongst patients from the intervention group. The anaesthetic interventions of interest are only those given to increase the mitoPO2 values. For all these interventions, we look for the difference between aggregated mitoPO2 values over a period before administering the anaesthetic intervention and aggregated mitoPO2 values over a period when the treatment is active. The lengths of the intervals, the time between intervals, and the type of aggregation are based on the observable patterns in the data. The time between intervals is at least the average time for the anaesthetic intervention to reach maximum plasma concentration; this duration may be longer because the effect could be delayed. If possible, we summarise the effect of the anaesthetic interventions by type and dose.
Effect when using the COMET in sequentially treated patients in mitoPO2 assessed with a mixed effects model | during surgery
  The relationship between the intervention number of patients from the interventions group sequentially treated by one anaesthetist and the mean intraoperative mitoPO2 value. The effect is defined as the average increase in mean intraoperative mitoPO2 when an anaesthetist treats a new patient from the intervention group.

OTHER OUTCOMES:
MitoPO2 for patients with epidural anaesthesia | during surgery
  Similair as the primary outcome, but exploring the effect in patients with or without epidural anaesthesia [2].
MitoPO2 for patients per surgical type | during surgery
  Similair as the primary outcome, but exploring the effect in patients with open versus laparoscopic surgical procedure [3].
MitoPO2 below 20 mmHg and 33 mmHg | during surgery
  The percentage of surgery time that the mitoPO2 is below 20mmHg and below 33 mmHg [4,5].

CONTACTS AND LOCATIONS:
Overall Officials: Markus W Hollmann, Professor, Principal Investigator — Amsterdam UMC, University of Amsterdam, Department of Anaesthesiology; Stijn W de Jonge, MD, Study Director — Amsterdam UMC, University of Amsterdam, Department of Surgery
Locations (1):
- Amsterdam UMC, University of Amsterdam, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kabon B, Fleischmann E, Treschan T, Taguchi A, Kapral S, Kurz A. Thoracic epidural anesthesia increases tissue oxygenation during major abdominal surgery. Anesth Analg. 2003 Dec;97(6):1812-1817. doi: 10.1213/01.ANE.0000087040.48267.54. PMID 14633566
- [Result] Fleischmann E, Kugener A, Kabon B, Kimberger O, Herbst F, Kurz A. Laparoscopic surgery impairs tissue oxygen tension more than open surgery. Br J Surg. 2007 Mar;94(3):362-8. doi: 10.1002/bjs.5569. PMID 17143850
- See also: Reference 1. Network NHS. Surgical Site Infection (SSI) Events — http://www.cdc.gov/nhsn/psc/ssi/index.html
- See also: Reference 4. de Wijs C, et al. MITOCHONDRIAL OXYGENATION DURING CARDIOPULMONARY BYPASS: A PILOT STUDY [abstract]. Virtual: In: EACTAIC-ICCVA Joint Congress / Journal of Cardiothoracic and Vascular Anesthesia 35 (2021) S1-S21, 2021 — http://www.eactaic.org/wp-content/uploads/2021/10/YJCAN_35_S1-1.pdf
- See also: Reference 5. Hilderink B, et al. Mitochondrial oxygen tension in patients after cardiac surgery: preliminary results [abstract]. Madrid, Spain: In: European society of intensive medicine LIVES 40, 2022 — http://esicmlives40.process.y-congress.com/ScientificProcess/schedule/?sessionGuid=0e0f17ea-3753-4e89-b3a5-d13e124a6e7b